CLINICAL TRIAL: NCT02215785
Title: Improvement of Functional Constipation With Kiwifruit Intake in a Mediterranean Patient Population: Open Non-controlled and Non-randomized Longitudinal Study
Brief Title: The Effect of Consumption of Kiwifruit on Constipation in Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 4R13/055
Record Dates: First submitted 2014-08-12; First posted 2014-08-13 (Estimated); Last update posted 2014-08-13 (Estimated); Status verified 2014-08

CONDITIONS: Constipation
Keywords: Funtional constipation; Kiwifruit; Health promotion
MeSH Terms: conditions — Constipation | interventions — alcohol acyltransferase, Actinidia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- kiwifruit cohort (Experimental): Patients that presented at Primary Care Centres with registered -Roma III criteria based- constipation and who accepted to participate in the study were followed-up for two weeks before intervention and three weeks under 3-daily kiwifruit intake.
  Interventions: Other: Kiwifruit

INTERVENTIONS:
Other: Kiwifruit — Throughout the five-week study period the patient had to continue their normal eating habits and exercise regime.
  Other Names: Green kiwifruits (Actinidia deliciosa var Hayward)

SUMMARY:
Constipation is a symptom suffered by a large number of people, due to multifactorial causes. Some studies have proven that modifying lifestyle reduces the risk of constipation, with high-fibre diets being less prone to constipation. Kiwifruit consumption, improves functional constipation and some studies consistently report an increase in the frequency and ease of defecation, stool volume and softness.

Although literature suggests kiwifruit consumption improves constipation symptoms, no studies have been carried out in adults and in Mediterranean patient populations, characteristic for its differential nutritional habits. The aim of the present study was to test the effect of kiwifruit consumption on functional constipation in a Spanish adult population.

DETAILED DESCRIPTION:
Worldwide general population prevalence of constipation ranges from 0.7% to 79% (median 16%). Some factors associated with constipation are sex, with higher prevalence in females (especially during pregnancy, and age; in general it becomes gradually more prevalent after the 70 years of age, in women the increase is considerable from a young age (18-23 years old) to middle age (45-50 years old).

Constipation is characterized by difficult or infrequent deposition, often accompanied by excessive straining during bowel movement or sensation of incomplete evacuation. In most cases, there is no underlying organic cause, and constipation is labelled as chronic idiopathic constipation and as a functional digestive disorder. The Rome III criteria is a useful tool for the diagnosis of constipation that highlights the chronic nature of the disorder and the importance of symptoms beyond the infrequency of bowel movements.

Understanding its causes, prevention, and treatment will help most people find constipation relief. An individual's medical history is very important in determining a constipation diagnosis. Primary healthcare professionals should enquire about dietary habits and lifestyle, pharmacological and toxic habits, complementary and alternative medicine, physiological bowel habits, use of laxatives and past disease history

Aims:

To test the effect of kiwifruit consumption on functional constipation in a Spanish adult population

Methods:

Design :Open non-controlled and non-randomized longitudinal study, of the effect of kiwifruit consumption in adult patients with diagnosed constipation

Setting: The study was conducted in five primary healthcare centres in Barcelona, Catalonia, Spain.

Period Study: Between April and August 2013

Population: Fifteen participating Primary Care Professionals selected patients from the electronic medical records (e-HCAP) following inclusion and exclusion criteria. Each professional could include a maximum of 4 patients. Forty-six subjects were selected for the study

Sample size: It was calculated to detect a change in the proportion of individuals with 3 or more defecations per week from 56% to 86% (evolution from an average of 3.2 to 4.4 -stable Standard Deviation (SD) of 1.3- in a normal distribution). Assuming a bilateral contrast for paired data, with a significance level of 0.05 and power of 0.8, a sample of 44 individuals was required (covering a 10% of dropout rate).

Intervention: The duration of the study was five weeks. During the first two weeks no kiwifruit patients were asked to follow their normal diet. The next three weeks they were asked to consume three Zespri green kiwifruits (Actinidia deliciosa var Hayward) per day, one at each main meal (breakfast, lunch and dinner). Throughout the five-week study period the patient had to continue their normal eating habits and exercise regime.

Tools and instructions: Primary Care Professionals asked patients to participate in the study and explained it to them. Patients who voluntarily agreed to participate signed the informed consent, accepting all study procedures. Each participant in the study attended three consultations: the first one before starting the study, the second one after two weeks and the third one after five weeks.

To collect the information patients used a questionnaire designed for this purpose. His/her Primary Care Professional provided instructions on the recording of faecal characteristics. The French original version of the diary was translated into Spanish and Catalan. Patients chose their own language to respond. Professionals collected data from diaries in a Google Docs form.

Patients were supplied kiwifruits in a heterogeneous manner. Some patients in the study bought the prescribed product. In other cases it was the professional who provided the kiwifruits. In one of the Primary Care Centres, the neighbourhood shopkeeper was the responsible for delivering the kiwifruits to the patients. Patients who bought their own Zespri kiwifruit were refunded.

Statistical analysis: Demographics for patients were summarized calculating medians [InterQuartile Range (IQR)] for continuous variables and proportions for categorical variables. Categorical variables were compared from baseline (second week) to last week using the Bhapkar test. For some analyses, Facility and Volume categorical variables were treated as continuous in order to provide results easy to interpret and taking into account individuals' correlations; in these cases, one unit of gain should be interpreted as an improvement in one response category. Functional data methodology was used for some graphical representations. Stacked barplots over time will be presented for categorical variables. To analyse week changes in daily variables Generalized Estimating Equation (GEE) models were adjusted (treating variables as continuous).

ELIGIBILITY:
Inclusion Criteria:

* Two or more of the following:

Straining during at least 25% of defecations Lumpy or hard stools in at least 25% of defecations Sensation of incomplete evacuation for at least 25% of defecations Sensation of anorectal obstruction/blockage for at least 25% of defecations Manual manoeuvres to facilitate at least 25% of defecations (e.g., digital evacuations and support of the pelvic floor) Fewer than three defecations per week; and

* Loose stools are rarely present without the use of laxatives;
* Insufficient criteria for irritable bowel syndrome;
* Criteria fulfilled for at least 3 months with symptom onset at least 6 months before diagnosis.

Exclusion Criteria:

* Patients with allergy to kiwifruit or latex
* Patients who have undergone gastro-intestinal surgery in the last year
* Patients taking medication to treat constipation
* Patients with oncological disease
* Patients taking narcotic medication
* Patients with organic gastroenterological diseases (except non- complicated diverticulosis).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2013-04; Primary Completion 2013-08 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with three or more stools per week | Five weeks
  Number of patients with three or more stools among participants Number of diary depositions recorded in a self adminitered questionnaire designed for this purpose
Frequency of stool per week | Five weeks
  Number of diary depositions recorded in a self adminitered questionnaire designed for this purpose
Number of responders (increase of ≥ 1 stool per week) | Five weeks
  Number of people increasing more ≥ 1stool for week recorded in a self adminitered questionnaire designed for this purpose

SECONDARY OUTCOMES:
Consistency of stool | Five weeks
  Bristol Scale: classified as Type 1 (Separate hard lumps, like nuts -hard to pass), Type 2 (Sausage-shaped, but lumpy), Type 3 (Like a sausage but with cracks on its surface), Type 4 (Like a sausage or snake, smooth and soft), Type 5 (Soft blobs with clear cut edges -passed easily-), Type 6 (Fluffy pieces with ragged edges, a mushy stool), or Type 7 (Watery, no solid pieces. Entirely liquid).
Volume of stool | Five weeks
  Classified as: very little (1), little (2), medium (3), reasonably much (4), a lot (5).
Ease of defecation | Five weeks
  Classified as: very easy (1), easy (2), normal (3), difficult (4), very difficult (5).
Satisfaction of the patient. | Five weeks
  Patients answer eight questions related to the improvement of defecation habits and quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Marta Besa Castellà, Dr, Study Chair — Catalan Institute of Health (ICS); Francisco Berlanga López, Study Chair — Catalan Institute of Health (ICS); Caterina Calvet Torres, Dr, Study Chair — Catalan Institut of Health (ICS); M Àngeles Cisneros Antó, Study Chair — Catalan Institut of Health (ICS); Judith Company Fontané, Study Chair — Catalan Institut of Health (ICS); Rosa Ma Clofent Vilaplana, Dr and Ph.D, Study Chair — Catalan Institut of Health (ICS); Caridad Delgado López, Dr, Study Chair — Catalan Institu of Health (ICS); Ma Isabel Denche Naranjo, Study Chair — Catalan Institut of Health (ICS); Maite Escudero Ruiz, Study Chair — Catalan Institut of Health (ICS); Angela Ferreres Castell, Study Chair — Catalan Institut of Health (ICS); Sonia Fuentes Rodriguez, Dr, Study Chair — Catalan Institut of Health (ICS); Amparo Gallart Iglesias, Study Chair — Catalan Institut of Health (ICS); M Roser Garriga Bacardí, Dr, Study Chair — Catalan Institut of Health (ICS); Isabel Marin Quilez, Study Chair — Catalan Institut of Health (ICS); Mercè Marzo Castillejo,, Dr and Ph.D, Principal Investigator — Catalan Institut of Health (ICS) and IDIAP Jordi Gol; Juanjo Mascort Roca, Dr, Study Chair — Catalan Institut of Health (ICS); Maria Ollé Mitjans, Dr, Study Chair — Catalan Institut of Health (ICS); Vanesa Pérez Martín, Study Chair — Catalan Institut of Health (ICS); Francesca Peñas López, Dr, Study Chair — Catalan Institut of Health (ICS); Gemma Nerin Pueyo, Study Chair — Catalan Institut of Health (ICS); Rosa Ramírez Torralbo, Dr, Study Chair — Catalan Institut of Health (ICS); Mercedes Rodriguez Pascual, Study Chair — Catalan Institut of Health (ICS); Laura Ruipérez Martín, Study Chair — Catalan Institut of Health (ICS); Josefa Ruiz Tejero, Study Chair — Catalan Institut of Health (ICS); Sonia Varela Folgueiras, Study Chair — Catalan Institut of Health (ICS); Carmen Vela Vallespín, Dr, Study Chair — Catalan Institut of Health (ICS); Mercè Vilarrubi Estrella, Dr, Study Chair — Catalan Institut of Health (ICS); Ivan Villar Balboa, Dr, Study Chair — Catalan Institut of Health (ICS)
Locations (1):
- Jordi Gol Gurina Foundation, Barcelona, Catalonia, Spain